CLINICAL TRIAL: NCT02396069
Title: A Phase I Clinical Study, Randomized, Double-blind, Placebo-controlled, Multiple Doses, Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics/Pharmacodynamics of JPI-289 in Healthy Male Volunteers.
Brief Title: The Evaluation of Safety, Tolerability and Pharmacokinetics/Pharmacodynamics of JPI-289 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JP-NC-P1-14
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2015-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — JPI-289

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JPI-289 (Experimental): Each cohort, volunteers will be infused JPI-289 for 60 min. (6 volunteers per each cohort, total 3 cohort)
  Interventions: Drug: JPI-289
- Placebo (Placebo Comparator): Each cohort, volunteer will be infused placebo for 60 min. (2 volunteers per each cohort, total 3 cohort)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JPI-289 — PARP-1 inhibitor
  Arms: JPI-289
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Double blind, randomized, placebo control, multiple dose, dose escalation study

DETAILED DESCRIPTION:
A phase I clinical study, randomized, double-blind, placebo-controlled, multiple doses, dose escalation study of the safety, tolerability and pharmacokinetics/pharmacodynamics of JPI-289 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 19~55 years healthy male
* BMI measurement 20kg/m²~27kg/m²
* 90 ≤ SBP<140(mmHg) 60 ≤ DBP<100(mmHg) 45 ≤ Pulse rate<100(bpm)
* Signed the informed consent form to participate voluntarily and to comply with the trial requirements
* For a follow-up visit and during the study period, blood samples and availability

Exclusion Criteria:

* History of clinically significant hepatic, gastrointestinal, pulmonary, musculoskeletal, endocrine, psychiatric, hematooncologic, cardiovascular (Specially asthma, obstructive pulmonary disease, peptic ulcer)
* History of skin disease of graft affecting absorption of the drug
* History of drug abuse
* Positive urine drug screening
* Administrated investigational product in a previous clinical trial within 60 days of the screening test
* Donated blood within 60 days prior to screening test

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss and Cmax,ss(76h), Relative PAR level(73h,%) | 96 hours, 73 hours

SECONDARY OUTCOMES:
Cav,ss | 96 hours
t1/2β | 96 hours
Vd,ss | 96 hours
CL | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No